CLINICAL TRIAL: NCT05385484
Title: A Savings Intervention to Reduce Men's Engagement in HIV Risk Behaviors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Impact Research & Development Organization (Other); University of California, San Francisco (Other); University of Washington (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 849897; 1R01HD103563-01A1 (NIH)
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus; STI; Alcohol Consumption; Incentives; Behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Alcohol Drinking; Behavior

STUDY DESIGN:
Intervention Model Description: In Kenyan communities with high HIV/STI prevalence, men will be randomized to two groups: a control group that receives basic health and financial education or a savings intervention group that receives a mobile banking account with incentives to save.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile banking account with incentives to save (Experimental): Participants in the savings intervention group will be provided with basic information on the importance of saving for the future, as well as (a) lottery-based incentives to save, (b) opportunities to develop savings goals, and (c) periodic reminders about the savings incentives and goals. Participants will receive assistance in opening and using a mobile savings account and will receive an education session that emphasizes the importance of saving for the future. Participants will be told about lottery-based incentives for saving money in their account.
  Interventions: Behavioral: Receives mobile banking account with incentives to save
- Basic health and financial education (No Intervention): Participants in the control group will be given basic information on the importance of saving for the future. In addition, health education curriculum developed by Impact Research & Development Organization (IRDO) will be provided to participants with standard health education on places to seek services for HIV and STI prevention and treatment, including information on alcohol and transactional sex as risk factors for HIV transmission.

INTERVENTIONS:
Behavioral: Receives mobile banking account with incentives to save — Participants will receive assistance in opening and using a mobile savings account, will be given education emphasizing saving practices and will be told about lottery-based incentives opportunities.
  Arms: Mobile banking account with incentives to save

SUMMARY:
This randomized control trial will test an economic intervention to reduce Kenyan men's engagement in behaviors that increase the risk of HIV/STIs. Participants randomized to the intervention group will be able to open accounts with a partner bank and will be incentivized to save with lottery-based rewards.

DETAILED DESCRIPTION:
This project will evaluate an innovative, theoretically-motivated economic intervention to reduce men's engagement in transactional sex and other risky behaviors. Leveraging innovations in mobile financial services and research on savings behavior in low-income countries, the investigators propose to test an intervention that seeks to motivate high-risk, income-earning men in western Kenya to reduce their spending on risky behaviors and instead save their disposable income in local bank accounts. These bank accounts will include additional incentives to save in the form of lottery-based rewards linked to amounts saved. The intervention will also encourage participants to develop savings goals and strategies, and provide periodic reminders about saving regularly. Through a direct economic mechanism (incentives to shift expenditures from the present to the future) and a psychological mechanism (increasing future orientation), the investigators hypothesize that the intervention will result in increased savings, reduced spending on transactional sex and alcohol, less risky sexual behavior, and reduced risk of HIV and sexually transmitted infections (STIs).

The investigators will conduct a randomized controlled trial among men who are at high risk of HIV and STI infection and determine the effects of a savings intervention on health and economic outcomes. Specific aims of the project are as follows. Aim 1: Determine the impact of the intervention on savings and investment behavior, self-reported sexual behavior, and incidence of HIV/STIs. Aim 2: Quantitatively and qualitatively assess mechanisms of behavior change among participants and a sample of their female partners.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-39 years
* Resides in study community and plans to remain for the next 2 years
* Used alcohol or other substances in the past month
* Engagement in any transactional sex (defined as payment of money, goods, or services in exchange for sex) in the past 3 months
* Has a steady income source that typically results in earnings every week
* Owns mobile phone
* Already has or is willing to open an account with partner banking institution
* Has national identification card (required for opening bank account)
* Has Kenya Revenue Authority personal identification number or is willing to create one (required for opening bank account)

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of HIV and other STIs | 24 months
  Composite incidence of at least one of HIV or other STIs (herpes simplex virus type 2 (HSV-2), Neisseria gonorrhoeae (NG), and Chlamydia trachomatis (CT)) over 24 months. The investigators will combine all STIs (including HIV) into a composite variable, with each participant counting once. For participants who are HIV-positive at baseline or HSV-2-positive, the outcome will be defined over all STIs other than HIV.

SECONDARY OUTCOMES:
Expenditures on alcohol (self only) | 6 month intervals
  Money spent on alcohol.
Expenditures on alcohol (self and others) | 6 month intervals
  Money spent on alcohol.
Expenditures on transactional sex | 6 month intervals
  Money, goods, and services spent on transactional sex (defined broadly to include financial and non-financial transfers to commercial and non-commercial sexual partners).
Expenditures on gambling | 6 month intervals
  Money spent on gambling.
Number of sexual partners | 6 month intervals
  Number of sexual partners participant had in the past 3 months.
Recent engagement in transactional sex | 6 month intervals
  Whether participant engaged in transactional sex (defined broadly to include financial and non-financial transfers to commercial and non-commercial sexual partners), or not in the past 3 months.
Number of transactional sex partners | 6 month intervals
  Total number of transactional sex partners participant had in the past 3 months.
Number of transactional sex encounters | 6 month intervals
  Number of transactional sex encounters participant engaged in during the past 3 months.
Condom use at most recent sexual encounter | 6 month intervals
  Whether participant used a condom or not at most recent sexual encounter in the past 3 months.
Alcohol use | 6 month intervals
  As measured by the Alcohol Use Disorders Identification Test-Concise (AUDIT-C) scale. The AUDIT-C is scored on a scale of 0-12, and higher values mean worse outcomes
HIV, CT, and NG incidence between 0-12 months and 12-24 months | Up to 24 months
  More temporally granular measures of incidence for HIV, CT, and NG.
Engagement in care among those who are HIV-positive | 6 month intervals
  Whether or not participants who are HIV-positive are currently engaged in care for their HIV.
Expenditures on food | 6 month intervals
  Money spent on food items.
Expenditures on household needs | 6 month intervals
  Money spent on household needs (including personal items; clothing and shoes; household items; utilities; and transport)
Savings and investment | 6 month intervals
  Total savings and investment, defined as the money value of formal and informal savings as well as investments in physical and human capital.
Total informal savings | 6 month intervals
  The sum of savings held outside of formal institutions, including savings groups and money saved at home or elsewhere
Total formal savings | 6 month intervals
  The sum of savings balances in all formal bank accounts.
Total household assets | 6 month intervals
  Value of all assets.
Expenditure on human capital investment | 6 month intervals
  Money spent on human capital investment (e.g., spending on children's education).
Any housing improvements | 6 month intervals
  Any improvement to house (yes/no)
Perpetuation Intimate partner violence | 6 month intervals
  Perpetuation of physical, psychological, or sexual IPV
Experienced Intimate partner violence | 6 month intervals
  Experienced physical, psychological, or sexual IPV
Perceived financial security | 6 month interval
  10 item scale by Fu 2020 World Development
Food security | 6 month interval
  3 item scale from Household Food Insecurity Access Scale. 0 to 9 with higher scores indicating higher food insecurity
Stress | 6 month interval
  Cohen's Perceived Stress Scale, PSS. 0 to 40 with higher scores indicating higher perceived stress
Stress, helplessness | 6 month interval
  Perceived helplessness score (subscale of PSS). 0 to 24 with higher scores indicating higher helplessness
Stress, self-efficacy | 6 month interval
  Perceived self-efficacy score (subscale of PSS). 0 to 16 with higher scores indicating higher self-efficacy
Future orientation | 6 month interval
  Assessed by a commonly-used scale that asks participants to make hypothetical choices between money received at two different times (e.g., 1,000 Shillings in 1 month vs. 1,100 Shillings in 2 months)
Future orientation, well being | 6 month interval
  Cantril scale which measures participant's well-being. 0 to 10 with higher scores indicating higher well being
Future orientation, longevity | 6 month interval
  11-point scale that assesses participant's expectations about their longevity. 0 to 10 with higher scores indicating higher expectations about longevity

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Impact Research and Development Organization, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egbe TI, Omollo OD, Wesonga JO, Bair EF, Chakrabarti A, Putt ME, Celum CL, Camlin CS, Napierala S, Agot K, Thirumurthy H. A savings intervention to reduce men's engagement in HIV risk behaviors: study protocol for a randomized controlled trial. Trials. 2022 Dec 16;23(1):1018. doi: 10.1186/s13063-022-06927-0. PMID 36527120

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT05385484/SAP_000.pdf